CLINICAL TRIAL: NCT02144142
Title: Phase 2 Study Evaluating the Kinetic Properties of an Autologous Microbiome Transplant in Adult Atopic Dermatitis Patients
Brief Title: Evaluation of the Kinetic Properties of an Autologous Microbiome Transplant in Adult Atopic Dermatitis Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This sub-study was not done because main study results reached significance.
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Richard Gallo, Chair, Division of Dermatology, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSD 131244.3
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Atopic Dermatitis; Eczema
Keywords: Microbiome; Atopic dermatitis; Eczema; Bacteriotherapy
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Moisturizer with each subject's own antimicrobial bacteria (Experimental): Each subject will have a moisturizer containing their own antimicrobial bacteria species spread over their arms in the clinic
  Interventions: Biological: Moisturizer with each subject's own antimicrobial bacteria

INTERVENTIONS:
Biological: Moisturizer with each subject's own antimicrobial bacteria
  Other Names: Autologous microbiome transplant cream

SUMMARY:
Unlike healthy control skin, the skin of patients with atopic dermatitis (AD) is frequently colonized by Staphylococcus aureus (S. aureus), putting these patients at increased risk of S. aureus skin infections. In addition, research in the investigator's lab has shown that these patients have fewer protective Staphylococcal species such as Staphylococcus epidermidis (S. epidermidis) that are known to produce antimicrobial peptides that play a role in protecting the skin from invading pathogens. In this study, the study team will attempt to decrease S. aureus colonization and increase colonization by protective Staph species in AD patients by first culturing the bacteria on subjects' lesional AD skin. The study team will selectively grow the subject's protective Staph colonies and place them into a moisturizer. The first part of the study will determine the half-life of the bacteria-containing moisturizer. The bacteria-containing moisturizer will be applied to a subject's arm, and the subject will return at four different time points over the next three days for skin swabs of the arm that will be used to determine the amount and type of bacteria on the arm at those time points. In the second part of the study, the subject will apply moisturizer containing his own antimicrobial bacteria to one of his arms for a total of 6 times at a frequency determined by the half-life, which will be computed at the end of the first part of this experiment. The subject will return prior to the 7th application time point for skin swabs of the arm to ensure that there are still viable bacteria from the moisturizer present on the arm. In the third part of the study, each subject will receive both moisturizer as well as moisturizer plus his own antimicrobial bacteria. The subject will apply the moisturizer to one arm and the moisturizer plus bacteria to the other arm daily for a total of 15 days. Subjects will return to the clinic every 5 days for skin swabs and clinical evaluations. If the moisturizer containing bacteria is able to decrease the S. aureus colonization on subject's arms, the study team hypothesizes that subjects will have improvement of their AD symptoms.

DETAILED DESCRIPTION:
This study will be conducted as three experiments in accordance with the three aims of the study. Participants will consent to all three of the study experiments separately, as each experiment will have a different consent form. While individual subjects are able to participate in all three sub-studies if they are eligible for all three, there is no requirement for subjects to participate in more than one of the sub-studies. A total of 10 subjects will be enrolled in Experiments 1 and 2, and approximately 14 subjects will be enrolled in Experiment 3. Given that only approximately 75-80% of AD patients are colonized by S. aureus, we expect to screen closer to 18-20 subjects to fulfill the inclusion criteria. Subjects that withdraw from the study will be replaced.

Experiment 1: Determination of the stability of transplanted bacteria on the skin surface over time

This first portion of the study (Experiment 1) will consist of 7 office visits (Screening, Culture, Treatment, and 3 Follow-up visits) and one phone call to relay eligibility information. All office visits will occur at the UCSD Dermatology Clinic. The exact procedures for each visit are discussed below.

Screening Visit (Visit 1, Day 0) Prior to beginning any study procedures, subjects will first be asked to review and sign the informed consent form. After obtaining informed consent, the inclusion/exclusion criteria will be reviewed. A brief medical history and physical exam will be performed in helping to assess whether the subject meets the required criteria for the study. Female subjects of child-bearing potential will take a urine pregnancy test in our office to ensure that they are not pregnant. Patients who meet the inclusion and exclusion criteria will then have a skin swab performed on the lesional atopic dermatitis skin in one of their antecubital fossae (Kong et al, 2012 showed that AD subjects colonized by S. aureus have resident S. aureus bacteria throughout their skin surface, therefore we expect one swab to be sufficient), as well as a nasal culture swab to detect the presence of S. aureus in the nares. This will conclude the screening visit. The total time for this visit will be approximately 30 minutes.

Subjects who do not meet the inclusion/exclusion criteria due to the application or use of prohibited medications within the timeframe noted will be considered screen-failures. Skin swabs of these patients will not be performed. These subjects may return for another screening visit after completing the necessary wash-out period (7 days for topical medications, 28 days for oral medications) if they are interested in doing so.

Phone (Day 3 +/- 1) Subjects will be notified via telephone within 3 business days whether or not their skin and nasal swabs grew S. aureus. Subjects with a skin culture positive for methicillin sensitive S. aureus (MSSA) will be enrolled in the study. A culture visit appointment will be schedule for these participants. Subjects will be excluded if they have any of the following: a negative S. aureus skin culture or a skin culture positive for methicillin-resistant S. aureus (MRSA). The total phone conversation should take approximately 5 minutes.

Culture Visit (Day 7 +/- 4) Eligible subjects will return for a culture visit within approximately a week of their screening visit. During this visit we will take four (4) culture swabs from the subject's non-lesional (no AD) skin on their upper arms. These culture swabs will be placed in tryptic soy broth (TSB) until processed in the lab, where they will be used to grow the subject's antimicrobial peptide-producing Staph species to use for the autologous microbiome transplant. Subjects will also receive a bar of Dove moisturizing soap, which they will be instructed to use whenever they shower until after the follow-up visit is complete. Subjects with a positive S. aureus nasal culture at the screening visit (Visit 1) will also receive a tube of mupirocin ointment. They will be instructed on the application of mupirocin to the anterior nares bilaterally twice a day starting 5 days prior to their treatment visit. The total visit will take approximately 10 minutes.

Treatment Visit (Day 28 +/- 7) Eligible subjects with + S. aureus screening cultures will be enrolled in the study and instructed to return to the clinic approximately 28 days after their screening visit. This 3-week waiting period will allow laboratory staff to grow and prepare the subject's endogenous AMP-producing bacteria to be mixed with Cetaphil for application at the treatment visit. To simulate real-life scenarios as much as possible, the subject will be allowed to continue their usual activities during this study, including bathing, showering, and exercising. This visit will begin by reviewing the subject's interim medical history, including medication history to ensure that he/she did not use any topical AD treatments on their arms within 7 days or oral AD treatments within 28 days of this visit. For subjects who had a S. aureus (+) nasal culture at screening visit, a repeat nasal culture will be performed. For all subjects, a focused physical exam will then be performed of the subject's bilateral arms to ensure that there is no evidence of cracks, breaks or infections of the skin on the arms. Next we will pre-treat both of the arms with a regimen of washing with Dial liquid antibacterial soap, followed by wiping the arm with sterile gauze soaked with 70%, then 80% alcohol. Once the alcohol has dried, a thin coat of the subject's individualized AMT cream will then be applied to each arm by the gloved hands of a study coordinator. Five minutes after applying the cream, a quantitative washing will be performed on eczematous skin of one antecubital fossae, as well as on a non-lesional area of skin on the same arm. For each wash, a sterile stainless steel cylinder with an approximate area of 3.5 cm2 will be held firmly to the skin surface, and 2.5 mL of a sterile stripping fluid (SSFN) will be carefully instilled into the cylinder. The skin will then be massaged for 60 seconds using a sterile rubber policeman. The SSFN will be aspirated with a pipette and transferred to a sterile test tube. This entire process will be repeated a second time at the same site and the fluid pooled together. The pooled fluid will be analyzed in the lab via colony counting methods to determine the number of viable bacteria colonies on the skin surface. A skin swab of both lesional and non-lesional skin will then be taken. This will conclude the treatment visit. We expect this visit to take approximately 30 minutes.

Follow-up Visits During follow-up visits, each subject will return to the clinic for a quantitative wash of their lesional and non-lesional skin and a skin swab of their lesional and non-lesional skin. The 10 enrolled subjects will be divided into two groups, and each group will return for follow-up at different time points. The first five patients to enroll will be assigned to the first group, which will return for follow-up at the following time points: 1, 4, 8 and 24-hours after the transplant. The next five patients to enroll will be assigned to the second group, and will return for follow-up at these time points: 1, 2, 4 and 7 days after the transplant. The quantitative wash at the final follow-up time point will conclude the study for that participant. Each follow-up visit will take approximately 20 minutes.

The average survival of the transplanted Staph species on both lesional and non-lesional skin will be plotted for each time point. From this data we will be able to calculate the rate of decline of the bacteria after being transplanted, which will provide us with the bacteria's half-life.

Experiment 2: To establish the steady-state abundance of autologous microbiome transplant cream application necessary to achieve a density of transplanted bacteria similar to the average concentration of microbes on normal skin, approximately 105/cm2

Experiment 2 will consist of 4 office visits (Screening, Culture, Treatment, and Follow-up), as well as one phone call to relay eligibility information. All office visits will occur at the UCSD Dermatology Clinic. Subjects who are participating in both Experiment 1 and 2 must wait at least a period of time equivalent to 10 half-lives of the AMT cream before beginning the study procedures of Experiment 2. The Screening, Phone Call, and Culture Visits for Experiment 3 are the same as for Experiment 1. The Treatment Visit and Follow-Up Visits differ slightly from those in Experiment 1 and will be described below, with changes underlined.

Treatment Visit (Day 28 +/- 7) Eligible subjects with + S. aureus screening cultures will be enrolled in the study and instructed to return to the clinic approximately 28 days after their screening visit for the treatment visit. This 3-week waiting period between the culture and treatment visits will allow laboratory staff to grow and prepare the subject's endogenous AMP-producing bacteria to be mixed with Cetaphil for application at the treatment visit. To simulate real-life scenarios as much as possible, the subject will be allowed to continue their usual activities during this study, including bathing, showering, and exercising. This visit will begin by reviewing the subject's interim medical history, including medication history to ensure that he/she did not use any topical AD treatments on their arms within 7 days or oral AD treatments within 28 days of this visit. For subjects who had a S. aureus (+) nasal culture at screening visit, a repeat nasal culture will be performed. For all subjects, a focused physical exam will then be performed of the subject's bilateral arms to ensure that there is no evidence of cracks, breaks or infections of the skin on the arms. Next we will pre-treat one arm with a regimen of washing with Dial liquid antibacterial soap, followed by wiping the arm with 70% followed by 80% alcohol using sterile gauze. Once the alcohol has dried, a thin coat of the subject's individualized AMT cream will then be applied to one of the subject's arms by the gloved hands of a study coordinator. Five minutes later, a quantitative washing will be performed on eczematous skin of the antecubital fossae of the arm treated with the AMT cream, as well as on an area of non-lesional skin on this same arm. For each wash, a sterile stainless steel cylinder with an approximate area of 3.5 cm2 will be held firmly to the skin surface, and 2.5 mL of a sterile stripping fluid (SSFN) will be carefully instilled into the cylinder. The skin will then be massaged for 60 seconds using a sterile rubber policeman. The SSFN will be aspirated with a pipette and transferred to a sterile test tube. This entire process will be repeated a second time and the fluid pooled together. The pooled fluid will be analyzed in the lab via PCR to determine how many and what type of bacteria are present. A skin swab of lesional and non-lesional skin will also be completed. Subjects will then be given single-use aliquots of their own AMT cream and gloves to take home with them. They will be instructed to apply one of the aliquots to the same arm it was applied to during the treatment visit at a dosing interval determined based on the half-life calculated from the results of Experiment 1 for a total of 6 doses (the dose schedule predicted to achieve steady state). They will be instructed to wash their hands and put on gloves prior to each application of the cream. This will conclude the treatment visit. We expect this visit to take approximately 30 minutes.

Follow-up Visit (To occur at the time of the 7th application of the AMT cream) During the follow-up visit, subjects will return to the clinic for a quantitative wash of their lesional and non-lesional skin to determine the abundance of S. aureus at this visit. A skin swab of lesional and non-lesional skin will also be performed. This visit will conclude Experiment 2. It will last approximately 15 minutes.

Additional considerations: In this experiment, our goal is to establish the steady-state abundance of AMT using a bacterial density similar to the average concentration of microbes on normal skin, approximately 105/cm2. Using the results of Experiment 1, we can estimate the half-life of the bacteria on subject skin surface. It is possible that the AMT cream half-life as determined in Experiment 1 will be short, possibly even as short as a few hours. If the AMT cream does show a rapid loss of transplanted bacteria such that it is impractical to further increase the frequency of application of the AMT (assumed as greater than TID), and the dose of the AMT cannot be practically increased from standard 108 bacteria/gm, applied at 10 gm/m2, the subject will apply the maximal practical dose (109 bacteria/gm at 40gm/m2 ) at the maximal practical frequency (TID), and we will do this for one week to determine how many bacteria are present after this treatment approach. Although this is not likely from the data of Costello et al. in 2009, we want to have this back-up plan in place to allow the study to move forward. Although these results would not represent a steady-state, the data would be sufficient to enable design of a subsequent clinical trial or to conclude that a long term application approach is not worth further analyses.

Experiment 3: To measure the steady-state abundance of S. aureus on participant's skin

Experiment 3 will consist of 6 office visits (Screening, Culture, Treatment, and 3 Follow-up visits), as well as one phone call to relay eligibility information. All office visits will occur at the UCSD Dermatology Clinic. Subjects who have participated in Experiment 2 must wait at least a period of time equivalent to 10 half-lives of the AMT cream before beginning the study procedures of Experiment 3. The Screening, Phone Call, and Culture Visits for Experiment 3 are the same as for Experiment 1. The Treatment Visit and Follow-Up Visits differ slightly from those in Experiment 1 and will be described below, with changes underlined.

Treatment Visit (Day 28 +/- 7) Eligible subjects with + S. aureus screening cultures will be enrolled in the study and instructed to return to the clinic approximately 28 days after their screening visit. This 3-week waiting period will allow laboratory staff to grow and prepare the subject's endogenous AMP-producing bacteria to be mixed with Cetaphil for application at the treatment visit. AMP-producing bacteria will also be screened to ensure that it is not pathogenic. To simulate real-life scenarios as much as possible, the subject will be allowed to continue their usual activities during this study, including bathing, showering, and exercising. This visit will begin by reviewing the subject's interim medical history, including medication history to ensure that he/she did not use any topical AD treatments on their arms within 7 days or oral AD treatments within 28 days of this visit. For subjects who had a S. aureus (+) nasal culture at screening visit, a repeat nasal culture will be performed. For all subjects, a focused physical exam will then be performed of the subject's bilateral arms to ensure that there is no evidence of cracks, breaks or infections of the skin on the arms. The localized SCORAD and Eczema Severity Scale will be completed on each antecubital fossa. A TEWL meter will then be used to measure the TEWL of each antecubital fossa. Next we will pre-treat both arms with a regimen of washing with Dial liquid antibacterial soap, followed by wiping the arms with 70%, then 80% alcohol. Once the alcohol has dried, a thin coat of the subject's individualized AMT cream will then be applied to one arm by the gloved hands of a study coordinator, and Cetaphil lotion alone to the other arm. The two creams will be labeled as either 'Right' or 'Left' to allow the study to be conducted in a double-blind manner (both the subject and the clinical investigator/coordinator will be blinded as to which arm received which treatment). Five minutes later, a quantitative washing will be performed on eczematous skin of both antecubital fossae as well as on an area of non-lesional skin of both arms. For each wash, a sterile stainless steel cylinder with an approximate area of 3.5 cm2 will be held firmly to the skin surface, and 2.5 mL of a sterile stripping fluid (SSFN) will be carefully instilled into the cylinder. The skin will then be massaged for 60 seconds using a sterile rubber policeman. The SSFN will be aspirated with a pipette and transferred to a sterile test tube. This entire process will be repeated a second time and the fluid pooled together. The pooled fluid will be analyzed in the lab via colony counting methods to determine the amount of viable bacteria on the skin at this time point. Skin swabs of lesional and non-lesional skin of both arms will also be taken to determine what type and the abundance of each bacteria present on the skin. The subject will then receive single-use aliquots of his individualized AMT cream and Cetaphil lotion alone, as well as gloves, and instructed to apply one aliquot to its assigned arm at the dosing interval determined in Experiment 1 (but not to exceed TID). All aliquots will be labeled with either 'Left' or 'Right' depending on which arm they should be applied to based on whether the aliquot is of control Cetaphil lotion or the AMT cream. Since the two products are identical in appearance and consistency, subjects should not be able to distinguish between the two products. All subjects will be instructed to wash their hands and put on clean gloves before each aliquot application. This will conclude the treatment visit. We expect this visit to take approximately 60 minutes.

Follow-Up Visits 1, 2 and 3 (Days 33 +/- 2 days, 38 +/- 2 days, and 43 +/- 2 days respectively) Subjects will return to the clinic approximately every 5 days after the treatment visit for a follow-up visit. During this visit, any adverse reactions to the AMT cream will be recorded. Next, the localized SCORAD and Eczema Severity Scale will be used to score the severity of the subject's eczema on each of his antecubital fossae. The TEWL of each antecubital fossa will also be measured. Next, a quantitative wash will be performed on each arm in the region of the antecubital fossa as well as on an area of non-lesional skin on each arm. A skin swab of the lesional and non-lesional skin from both arms will then be performed. The subject will receive freshly prepared single-use aliquots of both the AMT cream and Cetaphil lotion labeled with either 'Left' or 'Right' depending on which arm the aliquot should be applied to (for follow-up visits 1 and 2 only). These activities will conclude the study visit and all study-related procedures. Each follow-up visit should take approximately 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who are not pregnant or lactating
* 18-80 years of age
* Diagnosis of atopic dermatitis for at least 6 months using the Hanifin and Rajka Diagnostic Criteria for atopic dermatitis
* Presence of lesional atopic dermatitis skin in both antecubital fossae
* Positive S. aureus colonization based on results of a skin culture taken from one of their AD-affected antecubital fossae during the screening visit

Exclusion Criteria:

* Use of any topical AD treatments (including topical steroids, topical calcineurin inhibitors) to either arm within one week of either screening visit
* Use of any oral/systemic AD therapies (antihistamines, steroids) within 28 days of either screening visit
* Severe AD that would worsen significantly from holding a participant's usual topical/oral AD medications for the time periods required in the inclusion/exclusion criteria (one week prior to the screening, treatment and follow-up visits for topical medications and 28 days prior to screening, treatment and follow-up visits and for oral medications)
* Subjects who have taken a bleach bath within a week prior to screening, or who take bleach baths during the study
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study
* Subjects with Netherton's syndrome or other genodermatoses that result in a defective epidermal barrier
* Any subject who is immunocompromised (e.g. provides researchers with a history lymphoma, HIV/AIDS, Wiskott-Aldrich Syndrome) or has a history of malignant disease (with the exception of non-melanomatous skin cancer). This information will be gathered verbally from the patient while taking a medical history from the patient, and will not involve further testing such as an HIV test.
* Subjects with a history of psychiatric disease or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol
* Active bacterial, viral or fungal skin infections
* Any noticeable breaks or cracks in the skin on either arm, including severely excoriated skin or skin with open or weeping wounds suggestive of an active infection or increased susceptibility to infection.
* Ongoing participation in another investigational trial
* Use of any oral or topical antibiotic for up to four weeks prior to screening
* Use of any systemic immunosuppressive therapy (e.g. cyclosporine, methotrexate, etc.) within four weeks of screening.
* Sensitivity to or difficulty tolerating Dove fragrance-free bar soap, Dial antibacterial liquid soap, Cetaphil lotion, or alcohol-based cleaners
* Known allergy to mupirocin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Survival of transplanted bacteria | 1 hour
  The amount of the subject's own antimicrobial Staph species that were transplanted onto the subject will be measured

SECONDARY OUTCOMES:
Survival of transplanted bacteria | 4 hours
  The amount of the subject's own antimicrobial Staph species that were transplanted onto the subject will be measured
Survival of transplanted bacteria | 8 hours
  The amount of the subject's own antimicrobial Staph species that were transplanted onto the subject will be measured
Survival of transplanted bacteria | 24 hours
  The amount of the subject's own antimicrobial Staph species that were transplanted onto the subject will be measured
Survival of transplanted bacteria | 48 hours
  The amount of the subject's own antimicrobial Staph species that were transplanted onto the subject will be measured
Survival of transplanted bacteria | 4 days
  The amount of the subject's own antimicrobial Staph species that were transplanted onto the subject will be measured
Survival of transplanted bacteria | 7 days
  The amount of the subject's own antimicrobial Staph species that were transplanted onto the subject will be measured

OTHER OUTCOMES:
Adverse events | 4 hours
  Any adverse reactions to the antimicrobial Staph-containing moisturizer will be recorded
Adverse events | 1 hour
  Any adverse reactions to the antimicrobial Staph-containing moisturizer will be recorded
Adverse events | 8 hours
  Any adverse reactions to the antimicrobial Staph-containing moisturizer will be recorded
Adverse events | 24 hours
  Any adverse reactions to the antimicrobial Staph-containing moisturizer will be recorded
Adverse events | 48 hours
  Any adverse reactions to the antimicrobial Staph-containing moisturizer will be recorded
Adverse events | 4 days
  Any adverse reactions to the antimicrobial Staph-containing moisturizer will be recorded
Adverse events | 7 days
  Any adverse reactions to the antimicrobial Staph-containing moisturizer will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Gallo, MD, PhD, Principal Investigator — University of California San Diego Division of Dermatology
Locations (1):
- University of California San Diego Dermatology Clinic, San Diego, California, United States